CLINICAL TRIAL: NCT04856956
Title: Testing Pediatric Rheumatology Diagnostic Decision Support in Clinical Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: PhenoSolve, LLC (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BCH.SC.02
Record Dates: First submitted 2021-03-17; First posted 2021-04-23 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Diagnostic Skills for Rheumatologic Conditions

STUDY DESIGN:
Intervention Model Description: This study is a parallel-design, randomized, controlled study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: No masking is possible for subjects, since they will know whether they are or are not using the software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Use of diagnostic decision support software) (Experimental): Trainee or nurse practitioner sees patient and uses diagnostic decision support software in developing their differential diagnosis and plan
  Interventions: Other: Diagnostic decision support software
- Control (Current process) (No Intervention): Trainee or nurse practitioner sees patient but doesn't use diagnostic decision support software in developing their differential diagnosis and plan

INTERVENTIONS:
Other: Diagnostic decision support software — Comparing use of decision support group (intervention group) to use only of common literature (control group) among pediatric trainees diagnosing patients with possible rheumatologic disorder
  Arms: Intervention (Use of diagnostic decision support software)

SUMMARY:
This study is designed to test the helpfulness of a diagnostic tool, SimulConsult, when clinicians are diagnosing pediatric rheumatic diseases. Trainees and nurse practitioners will use the software or not use it, and their differential diagnoses will be compared to those of attending physicians in the same clinical encounter, and then to definitive diagnoses weeks later after testing, if one is reached.

DETAILED DESCRIPTION:
The study aims to assess improvement in the clinical performance of trainees evaluating patients with a suspected rheumatologic disorder. The Intervention is the use of Diagnostic Decision Support Software (DDSS) already available as a Boston Children's Hospital resource.

* Main objective: To assess if the use of the DDSS by trainees and nurse practitioners can improve their diagnostic performance in developing a differential diagnosis and plan in real clinical use. (Studies have shown in prior research that the use of the DDSS does so for case vignettes, lowering diagnostic errors of trainees by 75%). The study will compare how closely the differential diagnosis and plan of the trainees and nurse practitioners approximate those of their senior Pediatric Rheumatology attending physician colleagues.
* Secondary objective: To assess how frequently the differential diagnosis of the trainees and nurse practitioners includes the definitive diagnosis by doing a manual chart review weeks after the visit. (Studies have shown in prior research that if the definitive diagnosis is in the initial differential diagnosis, the right tests get ordered, and diagnostic errors are avoided.)

The design is a parallel one, comparing subjects (trainees and nurse practitioners) using the DDSS (Intervention Arm) to subjects who do not use the DDSS (Control Arm). In both study arms, subjects may use all other traditional resources. Arm assignment will be by patient case rather than trainee / nurse practitioner to reduce variation due to each subject's different capabilities (years of training and familiarity with pediatric rheumatology).

ELIGIBILITY:
The subjects are trainees (rheumatology and rotating fellows) and nurse practitioners, not patients. The Attendings participate in their supervisory role, and their clinical judgments are recorded as a preliminary "gold standard", but they are not research subjects.

* Trainees seeing new pediatric patients with a potential rheumatologic disorder are eligible. They will be drawn from the pool of Rheumatology fellows (3), Allergy/Immunology fellows (6), rotating pediatric and occasional adult residents (1 - 2) per month)
* Nurse practitioners in Rheumatology (2).
* Rheumatology Attendings for these new patient visits will also be asked to participate but will be supervisory participants in the study, not subjects.

We anticipate 15 trainees plus nurse practitioners will participate. There are no exclusion criteria, and we do not anticipate screen failures; however, trainees and nurse practitioners may decline to participate for individual patients or the entire study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance against Gold Standard: Presence of Gold standard #1 diagnosis in trainee list | 1 day
  The study will compare the trainee's differential diagnosis and workup plan to those of the attending physician seeing the same patient. The Attending is considered at this stage as the "gold standard" and we aim to answer the question "how well does a trainee with a DDSS (and traditional resources) approximate an experienced, specialist Attending vs. a trainee with access only to more traditional resources?".

SECONDARY OUTCOMES:
Performance against definitive diagnosis: Presence of definitive diagnosis in trainee list | 6 weeks
  The study will do a manual chart review of the cases to find the definitive diagnosis (where available) to measure the frequency with which the definitive diagnosis was in the trainee's initial DDx.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Segal, MD PhD, Study Chair — PhenoSolve, LLC; Robert P Sundel, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be shared.
Supporting Information: CSR
Time Frame: 2021-2022

REFERENCES:
- [Background] Segal MM. Mobile medical computing driven by the complexity of neurologic diagnosis. J Child Neurol. 2006 Jul;21(7):595-9. doi: 10.1177/08830738060210071601. PMID 16970851
- [Background] Segal MM, Athreya B, Son MB, Tirosh I, Hausmann JS, Ang EY, Zurakowski D, Feldman LK, Sundel RP. Evidence-based decision support for pediatric rheumatology reduces diagnostic errors. Pediatr Rheumatol Online J. 2016 Dec 13;14(1):67. doi: 10.1186/s12969-016-0127-z. PMID 27964737
- [Background] Staffa SJ, Zurakowski D. Strategies in adjusting for multiple comparisons: A primer for pediatric surgeons. J Pediatr Surg. 2020 Sep;55(9):1699-1705. doi: 10.1016/j.jpedsurg.2020.01.003. Epub 2020 Jan 23. PMID 32029234
- [Background] Segal MM, Williams MS, Gropman AL, Torres AR, Forsyth R, Connolly AM, El-Hattab AW, Perlman SJ, Samanta D, Parikh S, Pavlakis SG, Feldman LK, Betensky RA, Gospe SM Jr. Evidence-based decision support for neurological diagnosis reduces errors and unnecessary workup. J Child Neurol. 2014 Apr;29(4):487-92. doi: 10.1177/0883073813483365. Epub 2013 Apr 10. PMID 23576414